CLINICAL TRIAL: NCT01180894
Title: A Multicenter, Randomized, Double-blind Comparison of Intravenous Iron Supplementation to Placebo for the Treatment of Anemia of Traumatic Critical Illness
Brief Title: IV Iron for the Anemia of Traumatic Critical Illness
Acronym: IATCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Trauma Research Institute (Other)
Responsible Party: Principal Investigator, Fredric Pieracci, Principal Investigator, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0705
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Trauma; ICU Anemia
Keywords: Trauma; Anemia; Iron; Erythropoeisis
MeSH Terms: conditions — Wounds and Injuries; Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron sucrose (Active Comparator): 100 mg IV TIW
  Interventions: Drug: Iron sucrose
- Placebo (Placebo Comparator): Pacebo - Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron sucrose — 100 mg IV TIW
  Other Names: Fe sucrose
  Arms: Iron sucrose
Drug: Placebo
  Other Names: control
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to determine whether intravenous iron supplementation of anemic, critically ill trauma patients improves anemia and reduces the need for a red blood cell transfusion.

DETAILED DESCRIPTION:
Nearly all trauma patients admitted to an intensive care unit (ICU) are anemic (low red blood cell counts). Anemia is an independent risk factor for poor outcomes, including infection, impaired wound healing, and death. Current therapies for ICU anemia are unsatisfactory: Red blood cell (RBC) transfusion is associated with an increased risk of immune suppression, infection, and organ failure. Furthermore, use of both hemoglobin replacement products and erythropoietin are limited by expense as well as unfavorable side effect profiles.

One principal cause of anemia in trauma ICU patients involves disturbances in iron metabolism. Iron is necessary to make RBCs, and a lack of iron delivered to the bone marrow results in anemia. Trauma causes diversion of iron from the bone marrow into storage, where it cannot participate in the generation of RBCs. This diversion of iron is caused by inflammatory proteins released as a result of tissue injury.

Previous work by the principal investigator among ICU patients suggested a benefit to oral iron supplementation administered in dosages similar to those used in a standard multivitamin. However, many patients were not able to tolerate oral medications, and this study was not specific to trauma patients. Additional research has suggested that intravenous iron supplementation is effective in treating anemic patients with other inflammatory conditions, such as cancer and inflammatory bowel disease. However, the benefit of intravenous iron supplementation has never been tested among anemic ICU patients, including trauma patients.

The current clinical trial will evaluate the risk/benefit profile of intravenous iron supplementation among anemic trauma ICU patients. The study will take place over several academic trauma centers with a long history of participation in translational research.

Anemia remains a devastating complication of trauma. Current treatment options are limited. Intravenous iron supplementation represents a targeted, cost-effective solution to this pervasive problem, the efficacy of which remains undefined.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission for trauma
* Adults (age ≥ 18 years)
* Anemia (hemoglobin < 12 g/dL)
* ≤ 72 hours from ICU admission
* Expected ICU length of stay ≥ 7 days

Exclusion Criteria:

* Active hemorrhage requiring RBC transfusion
* Iron overload (serum ferritin concentration ≥ 1,000 ng/mL) or any condition associated with iron overload (e.g., hemochromatosis, aceruloplasminemia
* Chronic inflammatory conditions (e.g., systemic lupus erythematosis, rheumatoid arthritis, ankylosing spondilitis)
* Pre-existing hematologic disorders (e.g., thalassemia, sickle cell disease, hemophilia, von Willibrand's disease, myeloproliferative disease)
* Macrocytic anemia (mean corpuscular volume ≥ 100 fL)
* Current use of immunosuppressive agents including corticosteroids (e.g., dexamethasone, hydrocortisone, methylprednisolone, prednisone, exclusive of inhaled corticosteroids), calcinurin inhibitors (e.g., cyclosporine, tacrolimus), antimetabolites (e.g., azathioprine), or biologics (e.g., OKT3, thymoglobulin)
* Use of recombinant human erythropoietin formulation within the prev 30 days
* Pregnancy or lactation
* Prohibition of RBC transfusion
* Stay of ≥ 48 hours duration in the ICU of a transferring hospital
* History of intolerance or hypersensitivity to either enteral or intravenous iron
* Moribund state in which death is imminent
* Enrollment in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD, MPH, Principal Investigator — Denver Health Medical Center, University of Colorado Health Science Center
Locations (6):
- United States (6):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - NewYork Presbyterian Medical Center/Weill Cornell Medical College, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Harborview Medical Center/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieracci FM, Stovall RT, Jaouen B, Rodil M, Cappa A, Burlew CC, Holena DN, Maier R, Berry S, Jurkovich J, Moore EE. A multicenter, randomized clinical trial of IV iron supplementation for anemia of traumatic critical illness*. Crit Care Med. 2014 Sep;42(9):2048-57. doi: 10.1097/CCM.0000000000000408. PMID 24797376
- See also: National Trauma Institute — http://www.nationaltraumainstitute.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (100 mg normal saline)
Period: Overall Study
Arm/Group | Iron Sucrose | Placebo
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
  100 mg Normal saline
- Total: Total of all reporting groups
Arm/Group | Iron Sucrose | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 56 | 66 | 122
  >=65 years | 13 | 5 | 18
Age, Continuous [Median (Full Range); unit: years] | 41.6 [18 to 83] | 40.4 [18 to 87] | 41.0 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 29 | 46
  Male | 58 | 46 | 104
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: RBC Transfusion
Description: The number of participants who underwent RBC transfusion.
Time Frame: 42 Days
Measure: Number; unit: participants
Groups:
- Placebo: Pacebo - Normal Saline
  Placebo
Arm/Group | Iron Sucrose | Placebo
Number analyzed (Participants) | 75 | 75
participants | 47 | 55

2. Secondary Outcome: Iron-deficient Erythropoeisis (IDE)
Description: An elevated eZPP is diagnostic of Iron-deficient erythropoiesis (IDE) and reflects the bone marrow iron supply regardless of total body iron.
Time Frame: 14 Days
Measure: Mean (Full Range); unit: micro mol: mol heme
Arm/Group | Iron Sucrose | Placebo
Number analyzed (Participants) | 30 | 27
micro mol: mol heme | 118 [64 to 344] | 118 [78 to 244]

3. Secondary Outcome: Infection
Description: The number of participants with at least one infection.
  Specific infections analyzed included VAP (Ventilator-Associated Pneumonia), bacteremia, and urinary tract infection (UTI).
Time Frame: 28 Days
Measure: Number; unit: participants
Arm/Group | Iron Sucrose | Placebo
Number analyzed (Participants) | 44 | 52
participants | 1 | 1

4. Secondary Outcome: The Number of Participants Who Died
Time Frame: 28 Days
Measure: Number; unit: participants
Arm/Group | Iron Sucrose | Placebo
Number analyzed (Participants) | 75 | 75
participants | 7 | 2

ADVERSE EVENTS:
Arm/Group | Iron Sucrose | Placebo
Serious Adverse Events (participants affected / at risk) | 7/75 | 2/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Sucrose (N=75) | Placebo (N=75)
Mortality (Investigations) | 7 (7) | 2 (2) — In hospital mortality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No